CLINICAL TRIAL: NCT05747092
Title: Is Pain Killer Cunsumption Dependent to Anxiety or Mucogingival Therapy?
Brief Title: Pain Killer, Anxiety and Mucogingival Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Leila Salhi, PhD,Head of clinic, department of Periodontology, buccal surgery and buccal implantology,, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: B7072021000061
Record Dates: First submitted 2023-01-27; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Anxiety and Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: group test free gingival graft group control connective tissue graft
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: free gingival graft for gingival recession (Active Comparator)
  Interventions: Procedure: gingival graft
- Test group: connective tissue graft for gingival recession (Experimental)
  Interventions: Procedure: gingival graft

INTERVENTIONS:
Procedure: gingival graft — investigators:
  Donor site:
  * tissue graft harvesting from the palate behind the palatal rugae .
  * placement of a palatine hemostatic plaque on the palate in order to reduce the risk of bleeding and to diminish the postoperative pain.
  Received site:
  * Control: the horizontal incision adjacent to the recession(s) and vertical incisions and split thickness flap. Placement of the graft on the recipient bed and suture.
  * Test :connective tissue graft using the " envelope/pouch " technique with two partial thickness incisions (deep and superficial). Placement of the graft inside the envelope

SUMMARY:
Is the pain killer consumption after gingival treatment related to the level of patient anxiety or to the type of therapy?

DETAILED DESCRIPTION:
Anxiety and depression (HAD) scale used could be reveal the level of the patient anxiety and/or depression before intervention.

Additionnaly the use of these specific questionnaires (7 items for anxiety, 7 items for depression) could reveal if the pain killer consumption after gingical treatment is dependant to the level of HAD or to the therapy .

This tool (HAD) could allows to recognize, before any (oral)surgery, profil with high risk and propose solution to decrease anxiety and/or depression before treatment.

ELIGIBILITY:
Inclusion Criteria:

* ASA type I and II subjects
* Localized Gingival Recessions
* Recessions Cairo RT I-II
* FMPS < 10%
* FMBS< 10%
* <10 cigs/ day
* No contra-indication against oral surgical interventions
* Patient is able to give inform consent

Exclusion Criteria:

* Infection (local or systemic). Each infection will be evaluated prior to study procedure for suitability. Patients with gingivitis or local infection (fracture, apical reaction) will undergo a dental treatment prior to his entrance to the study. In case of systemic infection, the evaluation will be based on medical anamneses, and if necessary will be referred to relevant medical tests.
* ASA type > II
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Smokers, ≳ 10 cigarettes per day
* Immunocompromised patients
* Uncontrolled diabetes
* Untreated periodontitis
* History of previous periodontal surgery (mucogingival or other) on the teeth to be included
* Presence of severe tooth malposition, rotation or significant version of the tooth to be treated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
pin killer consumption | two weeks
  the number of pain killer used after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- leila Salhi, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No